CLINICAL TRIAL: NCT02456168
Title: Development of a Novel Glutamate Receptor Ligand for PET Scans in Neuropsychiatric Systemic Lupus Erythematosus
Status: Completed | Type: Observational
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Meggan Mackay, MD, Associate Investigator, MD, Northwell Health
Other Study IDs: PET CNS5161
Record Dates: First submitted 2015-05-15; First posted 2015-05-28 (Estimated); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Lupus; SLE
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- SLE
- Healthy control

SUMMARY:
Cognitive impairment occurs in as many as 80% of lupus patients and affective disorders, depression and anxiety, are also common. Both of these problems contribute significantly to disease burden and disability. Associations between serum anti-NMDAR Aab and cognitive and behavioral changes in human SLE have remained controversial, however, elevated titers of these Aabs in cerebrospinal fluid (CSF) correlate with severe central nervous system manifestations, such as coma and psychosis. The aim is to study the progression of disease (cognitive and behavioral impairment) over a 2 year period in SLE subjects with neuropsychologic and behavioral testing and correlates of disease progression using resting FDG-PET and serum Anti-NMDAR Aab. The correlations between hippocampal hypermetabolism, Anti-NMDAR Aab and memory impairment observed in the cross-sectional studies will be validated by baseline measurements in the proposed studies.

DETAILED DESCRIPTION:
Neuropsychiatric lupus is comprised of numerous, complex central and peripheral nervous system symptoms whose pathophysiologic mechanisms remain poorly understood. Cross-reactive anti-dsDNA antibodies have been shown to bind NR2A/NR2B subunits of the N-methyl D-aspartate receptor (NMDAR) on neurons and synergize with glutamate in a concentration dependent manner to either modulate receptor function or cause an excitotoxic, non-inflammatory neuronal death. Mice immunized to express anti-NMDAR Aab demonstrate a causal relationship between anti-NMDAR Aab and persistent behavioral and cognitive neuropathology following compromise to the blood brain barrier (BBB) which is necessary for Aab access to the brain.

The investigators' previous cross-sectional FDG-PET studies of resting brain glucose metabolism demonstrate robust hypermetabolism in the hippocampus of SLE subjects that associates independently with serum Anti-NMDAR Aab titer and impaired memory. Moreover, the combination of hippocampus hypermetabolism and elevated serum titers of Anti-NMDAR Aab has a higher predictive value for memory impairment than either variable alone. These significant correlations must be tested in a longitudinal study to evaluate the utility of FDG-PET as a biomarker for Anti-NMDAR Aab-mediated brain damage. The proposed longitudinal studies will inform the investigators about correlates of cognitive and behavioral change over time using FDG-PET imaging (Aim 1). Additionally, the investigators will explore NMDAR biology with a novel PET ligand, [11C]-CNS5161, used to localize and quantify NMDAR activation (Aim 2) and explore the role of blood brain barrier (BBB) integrity in cognitive and behavioral impairment (Aim 3).

ELIGIBILITY:
Inclusion Criteria:

1. Must be ≥18 and ≤55 years of age.
2. Must fulfill the current American College of Rheumatology (ACR) revised criteria for the diagnosis of SLE.
3. Must be willing and able to sign informed consent.
4. Must have stable disease activity and medication doses for 8 weeks prior to screening.

Exclusion Criteria:

1. History of neurological diseases including head injury resulting in a loss of consciousness, strokes (secondary to hypertension, atherosclerosis, diabetes), seizures, toxic exposure, any difficulties at birth, mental retardation.
2. History of documented transient ischemic attacks within six months of screening.
3. Currently taking anti-convulsant medication.
4. Limited fluency with English that in the opinion of the investigator would limit the subject's performance on the ACR battery of cognitive tests or the N-back task chosen for the working memory task during the PET scan.
5. History of illicit drug use (cocaine, cannabis, heroin) that can result in altered cognition.
6. Increased disease activity within 8 weeks defined by an increase in SLEDAI by 3 points or more, exclusive of points from serologies.
7. Any increase in steroid dose or addition of disease modifying agents within 8 weeks.
8. Exceeding the weight limit on the MRI scanner.
9. Suffering from claustrophobia.
10. Have any of the following: cardiac pacemakers, auto defibrillators, neural stimulators, aneurysm clips, metallic prostheses, cochlear implants, any implanted devices (pumps, infusion devices, stents), permanent eye make-up, IUD's, shrapnel injuries.
11. Current use of anxiolytic, antidepressant or antipsychotic medications.
12. Pregnant and/or lactating women
13. A glomerular filtration rate less than ≤60 mL/min or any evidence of active renal disease from any cause that would put the subject at risk for increased toxicity from gadolinium contrast for the MRI study.
14. The presence of uncontrolled or severe hypertension, diabetes mellitus or liver disease that would increase the risk of increased toxicity from gadolinium contrast.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 24 lupus subjects will be recruited based on the following Inclusion/Exclusion criteria and serum anti-NMDAR antibody status. The investigators are not selecting for SLE patients known to have cognitive or psychiatric disturbances because attribution of these problems is very difficult given the confounding effects of medications, co-morbid disease, metabolic disturbances and infections. The investigators are interested in the effects of the anti-NMDAR Aab and will stratify lupus subject population on this variable. The PET and MRI imaging studies will be performed only during times of stable disease activity and medication use to avoid confounding influences of acute changes in disease activity and steroids/immunosuppressive medications. The 17 healthy control subjects should have no history of chronic illness and be on no prescribed medications other than oral contraception. Subjects older than age 55 will also be excluded to avoid confounding effects of age on cognitive testing.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2014-01-21 (Actual); Primary Completion 2020-10-28 (Actual); Study Completion 2020-10-28 (Actual)

PRIMARY OUTCOMES:
Changes in brain activity | hippocampal metabolism from baseline over the 2 years

SECONDARY OUTCOMES:
Use of PET ligand CNS 5161 tracer as an assessment and imaging biomarker for regional brain dysfunction | Specific activity of CNS5161, determined by the UV absorbance of the radioactive peak as compared with a standard curve of CNS5161 from baseline over the 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Meggan Mackay, MD, Principal Investigator — Northwell Health
Locations (1):
- The Feinstein Institute for Medical Research, Manhasset, New York, United States